CLINICAL TRIAL: NCT05367739
Title: A Real-world Observational Study on the Efficacy and Safety of Anti HER2 Therapy
Brief Title: Real World Study on the Efficacy and Safety of Anti-HER2 Therapy
Status: Completed | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Real-HER2
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-07

CONDITIONS: Breast Neoplasms; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anti HER2 therapy can improve the survival of HER2 positive patients and reduce mortality. The aim of the open-label, real-world study is to assess efficacy and safety of Anti-HER2 treatment drugs.

DETAILED DESCRIPTION:
About 30% of breast cancer is human epidermal growth factor receptor-2 (HER2) amplification or overexpression (i.e. HER2 positive). HER2 positive breast cancer is one of the indicators of poor prognosis because of its high risk of invasion and metastasis. Anti HER2 therapy can improve the survival of HER2 positive patients and reduce mortality. The aim of the open-label, real-world study is to assess efficacy and safety of Anti-HER2 treatment drugs including antibody drugs such as trastuzumab and pertuzumab, small-molecule tyrosine kinase inhibitors (TKIs) such as lapatinib, neratinib, and pyrotinib, and antibody-drug conjugates such as trastuzumab deruxtecan (DS-8201) and trastuzumab emtansine (T-DM1).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, voluntary consent and signed written informed consent.
* ECOG 0~2.
* Diagnosis of locally advanced (stage IIIB or IIIC) or metastatic (stage IV) breast cancer.
* At least one measurable disease lesion before treatment.
* Anticipated survival time is longer than three months.
* Pathological and IHC reports for ER, PR, HER2 and Ki67 are available.
* For women with fertility, the pregnancy test before administration was negative, and agreed to take appropriate measures to avoid pregnancy during the study treatment and at least half a year after the end of treatment
* There are traceable medical records during treatment.

Exclusion Criteria:

* Pregnant or lactating women. Active infection requiring systemic treatment。
* HIV positive
* Suffering from or suspected of suffering from central nervous system diseases.
* Serious heart disease.
* Pulmonary lymphatic involvement leads to pulmonary dysfunction and requires active treatment, including the use of oxygen
* The investigator considered that the patient was not suitable for in this study, with any other situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 positive breast cancer patients who plan to receive anti-HER2 therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date of randomization until the date at the end of the second treatment cycle (42 days)
  The total rate of CR+PR after the completion of two cycles of treatment.
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The survival time from the date of recruitment to the date of the first documented progression or date of death.
Adverse Events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  All adverse events [including adverse events (AE / SAE) and ADR (adverse drug reactions)] will be collected when known. The classification of adverse reactions shall refer to CTCAE5.0 in case of adverse events / reactions. In case of serious adverse events, the investigators must immediately take necessary treatment measures to protect the safety of subjects. All adverse events / reactions should be tracked and observed. If the adverse events have not recovered, the investigator shall continue to give necessary treatment, report and record, and deal with special cases according to the management opinions of relevant departments.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China